CLINICAL TRIAL: NCT06290674
Title: Effect of Extracorporeal Shockwave on Abdominal Adiposity and Lipid Profile in Obese Postmenopausal Women
Brief Title: Extracorporeal Shockwave on Abdominal Adiposity and Lipid Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amany Ezzat Abbass Ali, Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004043
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Obesity, Abdominal
MeSH Terms: conditions — Obesity, Abdominal | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Clinical randomized controlled study
Who Masked: Participant, Investigator
Masking Description: Double masking (Investigator and Participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (A) (ESWT) (Active Comparator): 30 participants will receive Extracorporeal Shockwave (one session per week for 6 weeks), in addition to a balanced low-calorie diet (1500 k/cal for 6 weeks).
  Interventions: Other: Extracorporeal Shockwave therapy; Other: Balanced low-calorie diet
- Control Group (B) (Placebo Comparator): 30 participant will receive Balanced low-calorie diet (1500 k/cal for 6 weeks), only.
  Interventions: Other: Balanced low-calorie diet

INTERVENTIONS:
Other: Extracorporeal Shockwave therapy — 2000 shots, 120mJ pulse energy setting, 3 bar pressure, and 15 Hz for 15 minute per session.
  Arms: Study Group (A) (ESWT)
Other: Balanced low-calorie diet — 1500 k/cal for 6 weeks

SUMMARY:
Almost postmenopausal women store significant extra visceral adipose tissue with unexplained mechanism, yet. Postmenopausal obese women with excess abdominal obesity have raised metabolic risk of numerous cardiovascular diseases, which negatively influence health policy concern. Therefore, actual need to recommend non-invasive approach that cover this lack of quantitative knowledge in clinical management of obese postmenopausal women.

DETAILED DESCRIPTION:
Postmenopausal women are usually troubled by increasing weight and waist circumference caused by obesity and androcidal fat redistribution. Abdominal adiposity, defined as a waist circumference ≥88cm in women, measured in the upright position, plus significant elevated lipid profile values. In postmenopausal women, a higher level of physical activity was associated with a more optimal body composition, including lower adiposity and higher lean mass. Management of abdominal obesity involves different techniques i.e., dietary management, exercise therapy, even lifestyle management, and pharmacological management, and surgical interventions. Extracorporeal shockwave provides cavitation phenomena that may facilitate better management of abdominal obesity. Thus, current study will be conducted to investigate effect of extracorporeal shockwave on abdominal adiposity and lipid profile in obese post-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Their age range 45-60 years old.
* Their body mass index range 30-35 kg/m square.
* Only, obese postmenopausal women with at least one year after stoppage of menses.

Exclusion Criteria:

* Receiving pharmacological treatment.
* Receiving any form of electrotherapy.
* Whom with metabolic, hematological or renal dysfunction.
* Whom have dermatological or cardiovascular or respiratory, digestive or rheumatic disorders.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Current study focuses on Obese Postmenopausal women, based on well-known associated abdominal obesity.
Enrollment: 60 (Actual)
Dates: Start 2022-09-11 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Waist/ hip ratio | Pretreatment and Posttreatment of six weeks study protocol.
  anthropometric outcome measure for abdominal adiposity
Skin fold caliper | Pretreatment and Posttreatment of six weeks study protocol.
  subcutaneous fat outcome measure

SECONDARY OUTCOMES:
Lipid profile | Pretreatment and Posttreatment of six weeks study protocol.
  Low-density lipoprotein, High-density lipoprotein, and triglyceride laboratory outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Azza B Nashed, PHD, Study Chair — Professor of Physical Therapy for Women's Health; Sherif S El-Shebeni, MSc., Study Director — Consultant of Obstetrics and Gynecology
Locations (1):
- Helwan General Hospital, Cairo, Helwan, Cairo Governate, Egypt

IPD SHARING:
Plan to Share IPD: No
Will Share whole raw data, therapeutic protocol details for future systematic review and/ or meta-analysis. wish to be valuable